CLINICAL TRIAL: NCT06708429
Title: Impact of Immune-surveillance on the Development of Colorectal Cancer in Patients With Lynch Syndrome
Brief Title: Lynch Syndrome X-Talk of Enteral Mucosa With Immune System
Acronym: LYNX-EYE
Status: Recruiting | Type: Observational
Sponsor: San Raffaele University (Other)
Responsible Party: Sponsor
Other Study IDs: LYNX EYE 2023
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Lynch Syndrome; Lynch Syndrome I; Lynch Syndrome II; Lynch Syndrome I (Site-specific Colonic Cancer); HNPCC; HNPCC Gene Mutation; Hereditary Cancer Syndrome; Hereditary Cancer; MLH1 Gene Mutation; MLH1 Gene Deletion+Duplication; MLH1 Loss of Expression; MLH1 Gene Inactivation; MSH2 Gene Mutation; MSH2 Gene Deletion+Duplication; MSH2 Loss of Expression; MSH2 Gene Inactivation; MSH6 Gene Mutation; MSH6 Loss of Expression; MSH6 Gene Inactivation; PMS2 Gene Mutation; PMS2 Gene Inactivation; PMS2 Loss of Expression
Keywords: Colorectal cancer; Endometrial cancer; Lynch syndrome-associated cancer; Surveillance; Cancer surveillance; Immune profile; Immune escape; Mismatch repair deficiency; Microbiota; Liquid biopsy; MicroRNA; Transcriptomic; Frame shift peptides; MLH1; MSH2; EpCAM; MSH6; PMS2; Hair matrix
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Lynch Syndrome II; Lynch syndrome I (site-specific colonic cancer); Neoplastic Syndromes, Hereditary; Colorectal Neoplasms; Endometrial Neoplasms; Turcot syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Formalin-fixed, paraffine embedded mucosal samples Formalin-fixed, paraffine embedded tumor samples Hair matrix Plasma Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (14):
- Lynch syndrome (MLH1), without colorectal cancer and without advanced adenomas: A cohort of individuals with a germline pathogenic variant in the MLH1 gene, that confers a diagnosis of Lynch syndrome, who are found to be cancer-free and adenoma-free at the time of colonoscopy evaluation
  Interventions: Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System)
- Lynch syndrome (MLH1), with colorectal cancer or advanced adenomas: A cohort of individuals with a germline pathogenic variant in the MLH1 gene, that confers a diagnosis of Lynch syndrome, who are found to have colorectal cancer or an adenoma at the time of colonoscopy evaluation
  Interventions: Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System)
- Lynch syndrome (MSH2), without colorectal cancer and without advanced adenomas: A cohort of individuals with a germline pathogenic variant in the MSH2 gene, that confers a diagnosis of Lynch syndrome, who are found to be cancer-free and adenoma-free at the time of colonoscopy evaluation
  Interventions: Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System)
- Lynch syndrome (MSH2), with colorectal cancer or advanced adenomas: A cohort of individuals with a germline pathogenic variant in the MSH2 gene, that confers a diagnosis of Lynch syndrome, who are found to have colorectal cancer or an adenoma at the time of colonoscopy evaluation
  Interventions: Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System)
- Lynch syndrome (MSH6, without colorectal cancer and without advanced adenomas: A cohort of individuals with a germline pathogenic variant in the MSH6 gene, that confers a diagnosis of Lynch syndrome, who are found to be cancer-free and adenoma-free at the time of colonoscopy evaluation
  Interventions: Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System)
- Lynch syndrome (MSH6), with colorectal cancer or advanced adenomas: A cohort of individuals with a germline pathogenic variant in the MSH6 gene, that confers a diagnosis of Lynch syndrome, who are found to have colorectal cancer or an adenoma at the time of colonoscopy evaluation
  Interventions: Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System)
- Lynch syndrome (PMS2), without colorectal cancer and without advanced adenomas: A cohort of individuals with a germline pathogenic variant in the PMS2 gene, that confers a diagnosis of Lynch syndrome, who are found to be cancer-free and adenoma-free at the time of colonoscopy evaluation
  Interventions: Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System)
- Lynch syndrome (PMS2), with colorectal cancer or advanced adenomas: A cohort of individuals with a germline pathogenic variant in the PMS2 gene, that confers a diagnosis of Lynch syndrome, who are found to have colorectal cancer or an adenoma at the time of colonoscopy evaluation
  Interventions: Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System)
- Lynch syndrome (MSH2, exon 8 deletion), without colorectal cancer and without advanced adenomas: A cohort of individuals with a germline pathogenic exon 8 deletion in the MSH2 gene, that confers a diagnosis of Lynch syndrome, who are found to be cancer-free and adenoma-free at the time of colonoscopy evaluation
  Interventions: Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System)
- Lynch syndrome (MSH2, exon 8 deletion), with colorectal cancer or advanced adenomas: A cohort of individuals with a germline pathogenic exon 8 deletion in the MSH2 gene, that confers a diagnosis of Lynch syndrome, who are found to have colorectal cancer or an adenoma at the time of colonoscopy evaluation
  Interventions: Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System)
- Non-Lynch syndrome, with colorectal cancer: A cohort of individuals without a germline pathogenic variant in any of the mismatch repair genes (MLH1, MSH2, MSH6, PMS2), who are found to have colorectal cancer at the time of colonoscopy evaluation
  Interventions: Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System)
- Non-Lynch syndrome, with high-risk adenomas: A cohort of individuals without a germline pathogenic variant in any of the mismatch repair genes (MLH1, MSH2, MSH6, PMS2), who are found to have high-risk adenomas at the time of colonoscopy evaluation
  Interventions: Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System)
- Non-Lynch syndrome, with low-risk adenomas: A cohort of individuals without a germline pathogenic variant in any of the mismatch repair genes (MLH1, MSH2, MSH6, PMS2), who are found to have low-risk adenomas at the time of colonoscopy evaluation
  Interventions: Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System)
- Non-Lynch syndrome, without colorectal cancer and without colorectal adenomas: A cohort of individuals without a germline pathogenic variant in any of the mismatch repair genes (MLH1, MSH2, MSH6, PMS2), who are found to be cancer-free and adenoma-free at the time of colonoscopy evaluation
  Interventions: Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System)

INTERVENTIONS:
Diagnostic Test: LYNX EYE (Lynch syndrome X-Talk of Enteral mucosa with Immune System) — A combination of blood-based, mucosal-based, and hair-based analyses that evaluate the presence and the expression of:
  * a set of microRNAs (blood)
  * antibodies anti-frame shift peptides (blood)
  * mucosal-resident bacteria (healthy mucosa and cancer)
  * environmental exposure to potential carcinogens (hair matrix)

SUMMARY:
Lynch syndrome (OMIM #120435) is the most common dominantly inherited colorectal cancer syndrome with an estimated prevalence of 1:270 individuals. It increases the lifetime risk of colorectal and endometrial cancer primarily, but it is associated with a high risk of other cancers (pancreas, stomach, ovarian, central nervous system, skin, among others). It is caused by a germline mutation in one of four DNA mismatch repair genes or a terminal deletion of the MSH2-adjacent gene EpCAM.

Despite adherence to cancer surveillance programs, many patients still develop colorectal cancer and endometrial cancer. The Prospective Lynch Syndrome Database (PLSD) suggests that more frequent surveillance intervals do not significantly improve cancer risk reduction. The PLSD also revealed that the incidence of colorectal cancer in MLH1 and MSH2 carriers was even higher than previously expected, reaching as high as 41-36% among MLH1 carriers, regardless of ethnic background. The development of colorectal cancer despite surveillance is an unresolved question. Therefore, there is an unmet need for effective cancer prevention strategies.

DETAILED DESCRIPTION:
The risk of developing colorectal cancer in individuals with Lynch syndrome remains high despite endoscopic surveillance.

In Lynch Syndrome, the cancer-formation process is characterized by the development of immunogenic neo-antigens in the mucosa. These neoantigens, called frame-shift peptides, can be recognized by the adaptive immune systems, and trigger the formation of antibodies against them (termed anti-frame-shift peptides antibodies). Anti-frame-shift peptide antibodies have been reported in some Lynch syndrome patients (defined dichotomously as the presence vs absence of anti-frame-shift peptide antibodies). This study hypothesizes that anti-frame-shift peptide antibodies represent an early biomarker of cancer development in Lynch syndrome. These anti-frame-shift peptide antibodies may be used to identify early patients at the highest risk of developing colorectal cancer. All studies on anti-frame-shift peptide antibodies have had a cross-sectional design, while a retro-prospective design would be desirable to understand the interaction between the mucosa and the mucosa-associated immune system. There is also limited evidence that individuals with Lynch syndrome develop mismatch repair-deficient crypts before colorectal cancer development. The development of interval colorectal cancers may require specific biological processes. Understanding the biological processes underlying these interval colorectal cancers would help define targets of innovative therapies to prevent colorectal cancer (including but not limited to chemoprevention strategies and cancer vaccines). The interactions between the mucosa immune surveillance and the colonic epithelium are the cornerstone to answer such questions. Finally, the development of gastric cancer via non-canonical pathways (non-Correa, non-HPylori) demands a better understanding of the pathogenesis in individuals with Lynch syndrome.

MicroRNA (miRNA) expression has been shown to have diagnostic, prognostic, and therapeutic potential. While they offer high detection sensitivity, the heterogeneity limits their detection accuracy. Exosomes are excreted by cancer cells and possess specific exosomal miRNA signatures. Since circulating cell-free miRNAs offer excellent sensitivity but may suffer from inadequate specificity, while exosomal miRNAs are highly tissue-specific but might lack sensitivity, a combination of these biomarkers could offer an optimal combination of sensitivity and specificity. 98.5% of the total DNA is non-coding regions with roles in gene regulation, alternative splicing, interaction with transcription factors, and sequences capable of moving around the genome and promoting carcinogenesis. The understanding of non-coding DNA seems to be important in cancer early diagnosis.

Lynch syndrome-associated colorectal cancers are high immunogenic lesions with abundant lymphocyte infiltration. This study aims to develop an extensive profile of the immunosuppressive and regulatory cellular population in blood and tumor sites to identify patients with higher risks of cancer development.

Recent data have demonstrated the presence of intratumor bacteria in both cancer and immune cells. Therefore, this study also aims to analyze in colonic biopsies from Lynch syndrome patients with- and without tumors the presence of microbiota as an early signature for carcinogenesis.

ELIGIBILITY:
Inclusion Criteria (for participants with Lynch syndrome):

* Age ≥18 years
* All sexes eligible
* Established diagnosis of Lynch syndrome performed as part of clinical practice, with a germline pathogenic/likely pathogenic variant in one of the following genes: MLH1, MSH2, MSH6, PMS2, and EpCAM
* Subjects with Lynch syndrome undergoing surveillance gastrointestinal endoscopy and/or surgery according to clinical practice
* Fertile patients (both males and females) are eligible
* Lactating women are eligible

Inclusion Criteria (for participants without Lynch syndrome):

* Age ≥18 years
* All sexes eligible
* Patients with sporadic colorectal lesions, including colorectal cancer and colorectal adenomas
* Healthy controls without colorectal cancer or adenomas undergoing lower gastrointestinal endoscopy for abdominal pain
* PREMM5 < 2.5 [PREMM5 is an online, free-to-use, clinical prediction algorithm that estimates the cumulative probability of an individual carrying a germline mutation in the mismatch repair genes responsible for Lynch syndrome].

Exclusion Criteria (for participants with or without Lynch syndrome):

* Age < 18 years;
* Diseases that are known to predispose to colorectal cancer (personal past or recent history of inflammatory bowel disease);
* Patients unable/unwilling to provide consent;
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients with and without Lynch syndrome, with and without colorectal cancer or colorectal adenomas.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2033-06-01 (Estimated); Study Completion 2034-06-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 year
  True positive rate: the probability of a positive test result, conditioned on the individual truly being positive

SECONDARY OUTCOMES:
Specificity | Through study completion, an average of 1 year
  True negative rate: the probability of a negative test result, conditioned on the individual truly being negative
Proportion of correct predictions (true positives and true negatives) among the total number of cases (i.e., accuracy) | Through study completion, an average of 1 year
  A measure of trueness: proportion of correct predictions (both true positives and true negatives) among the total number of cases examined
Prevalence of anti-frame-shift peptide antibodies positivity in blood sample | Through study completion, an average of 1 year
  The proportion of individuals who have detectable levels of antibodies against frame shift peptides in their blood, conditioned on the individual truly being positive
Tumor microbiome analysis | Through study completion, an average of 1 year
  A comprehensive analysis of the tumor microbiome to identify high-risk patients for colorectal cancer onset
Immuno-environmental tumor signature | Through study completion, an average of 1 year
  A comprehensive evaluation of the differential expression of immunosuppressive myeloid-related signatures in colorectal lesions compared to healthy mucosa of patients with Lynch syndrome.
  A comprehensive evaluation of the differential expression of immunosuppressive myeloid-related signatures in the blood of individuals with Lynch syndrome, with vs. without colorectal cancer
Exposure analysis | Through study completion, an average of 1 year
  A comprehensive evaluation of the environmental exposure analysis on the hair matrix of individuals with Lynch syndrome, with vs. without colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Martina Cavestro, MD, PhD, Principal Investigator — IRCCS San Raffaele Scientific Institute
Locations (5):
- Beckman Research Institute at City of Hope, Monrovia, California, United States
- Italy (4):
  - Gastronterology and Gastrointestinal Endoscopy Unit, IRCCS San Raffaele Hospital, Milan, Lombardy
  - Dipartimento di Chirurgia Oncologica e Dipartimento di Oncologia Sperimentale Istituto Nazionale Tumori, Milan, MI
  - Dipartimento di controllo qualità e rischio chimico biologico, AOOR Villa Sofia Cervello, Palermo, PM
  - Chirurgia Generale, Azienda Ospedaliero Universitaria di Cagliari, Cagliari

IPD SHARING:
Plan to Share IPD: Undecided
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data.

REFERENCES:
- [Background] Lynch HT, Snyder CL, Shaw TG, Heinen CD, Hitchins MP. Milestones of Lynch syndrome: 1895-2015. Nat Rev Cancer. 2015 Mar;15(3):181-94. doi: 10.1038/nrc3878. Epub 2015 Feb 12. PMID 25673086
- [Background] Win AK, Jenkins MA, Dowty JG, Antoniou AC, Lee A, Giles GG, Buchanan DD, Clendenning M, Rosty C, Ahnen DJ, Thibodeau SN, Casey G, Gallinger S, Le Marchand L, Haile RW, Potter JD, Zheng Y, Lindor NM, Newcomb PA, Hopper JL, MacInnis RJ. Prevalence and Penetrance of Major Genes and Polygenes for Colorectal Cancer. Cancer Epidemiol Biomarkers Prev. 2017 Mar;26(3):404-412. doi: 10.1158/1055-9965.EPI-16-0693. Epub 2016 Oct 31. PMID 27799157
- [Background] Haraldsdottir S, Rafnar T, Frankel WL, Einarsdottir S, Sigurdsson A, Hampel H, Snaebjornsson P, Masson G, Weng D, Arngrimsson R, Kehr B, Yilmaz A, Haraldsson S, Sulem P, Stefansson T, Shields PG, Sigurdsson F, Bekaii-Saab T, Moller PH, Steinarsdottir M, Alexiusdottir K, Hitchins M, Pritchard CC, de la Chapelle A, Jonasson JG, Goldberg RM, Stefansson K. Comprehensive population-wide analysis of Lynch syndrome in Iceland reveals founder mutations in MSH6 and PMS2. Nat Commun. 2017 May 3;8:14755. doi: 10.1038/ncomms14755. PMID 28466842
- [Background] Engel C, Vasen HF, Seppala T, Aretz S, Bigirwamungu-Bargeman M, de Boer SY, Bucksch K, Buttner R, Holinski-Feder E, Holzapfel S, Huneburg R, Jacobs MAJM, Jarvinen H, Kloor M, von Knebel Doeberitz M, Koornstra JJ, van Kouwen M, Langers AM, van de Meeberg PC, Morak M, Moslein G, Nagengast FM, Pylvanainen K, Rahner N, Renkonen-Sinisalo L, Sanduleanu S, Schackert HK, Schmiegel W, Schulmann K, Steinke-Lange V, Strassburg CP, Vecht J, Verhulst ML, de Vos Tot Nederveen Cappel W, Zachariae S, Mecklin JP, Loeffler M; German HNPCC Consortium, the Dutch Lynch Syndrome Collaborative Group, and the Finnish Lynch Syndrome Registry. No Difference in Colorectal Cancer Incidence or Stage at Detection by Colonoscopy Among 3 Countries With Different Lynch Syndrome Surveillance Policies. Gastroenterology. 2018 Nov;155(5):1400-1409.e2. doi: 10.1053/j.gastro.2018.07.030. Epub 2018 Jul 29. PMID 30063918
- [Background] Moller P, Seppala T, Bernstein I, Holinski-Feder E, Sala P, Evans DG, Lindblom A, Macrae F, Blanco I, Sijmons R, Jeffries J, Vasen H, Burn J, Nakken S, Hovig E, Rodland EA, Tharmaratnam K, de Vos Tot Nederveen Cappel WH, Hill J, Wijnen J, Green K, Lalloo F, Sunde L, Mints M, Bertario L, Pineda M, Navarro M, Morak M, Renkonen-Sinisalo L, Frayling IM, Plazzer JP, Pylvanainen K, Sampson JR, Capella G, Mecklin JP, Moslein G; Mallorca Group (http://mallorca-group.eu). Cancer incidence and survival in Lynch syndrome patients receiving colonoscopic and gynaecological surveillance: first report from the prospective Lynch syndrome database. Gut. 2017 Mar;66(3):464-472. doi: 10.1136/gutjnl-2015-309675. Epub 2015 Dec 9. PMID 26657901
- [Background] Seppala T, Pylvanainen K, Evans DG, Jarvinen H, Renkonen-Sinisalo L, Bernstein I, Holinski-Feder E, Sala P, Lindblom A, Macrae F, Blanco I, Sijmons R, Jeffries J, Vasen H, Burn J, Nakken S, Hovig E, Rodland EA, Tharmaratnam K, de Vos Tot Nederveen Cappel WH, Hill J, Wijnen J, Jenkins M, Genuardi M, Green K, Lalloo F, Sunde L, Mints M, Bertario L, Pineda M, Navarro M, Morak M, Frayling IM, Plazzer JP, Sampson JR, Capella G, Moslein G, Mecklin JP, Moller P; Mallorca Group. Colorectal cancer incidence in path_MLH1 carriers subjected to different follow-up protocols: a Prospective Lynch Syndrome Database report. Hered Cancer Clin Pract. 2017 Oct 10;15:18. doi: 10.1186/s13053-017-0078-5. eCollection 2017. PMID 29046738
- [Background] Mecklin JP, Aarnio M, Laara E, Kairaluoma MV, Pylvanainen K, Peltomaki P, Aaltonen LA, Jarvinen HJ. Development of colorectal tumors in colonoscopic surveillance in Lynch syndrome. Gastroenterology. 2007 Oct;133(4):1093-8. doi: 10.1053/j.gastro.2007.08.019. Epub 2007 Aug 14. PMID 17919485
- [Background] Vasen HF, Abdirahman M, Brohet R, Langers AM, Kleibeuker JH, van Kouwen M, Koornstra JJ, Boot H, Cats A, Dekker E, Sanduleanu S, Poley JW, Hardwick JC, de Vos Tot Nederveen Cappel WH, van der Meulen-de Jong AE, Tan TG, Jacobs MA, Mohamed FL, de Boer SY, van de Meeberg PC, Verhulst ML, Salemans JM, van Bentem N, Westerveld BD, Vecht J, Nagengast FM. One to 2-year surveillance intervals reduce risk of colorectal cancer in families with Lynch syndrome. Gastroenterology. 2010 Jun;138(7):2300-6. doi: 10.1053/j.gastro.2010.02.053. Epub 2010 Mar 2. PMID 20206180
- [Background] Jarvinen HJ, Aarnio M, Mustonen H, Aktan-Collan K, Aaltonen LA, Peltomaki P, De La Chapelle A, Mecklin JP. Controlled 15-year trial on screening for colorectal cancer in families with hereditary nonpolyposis colorectal cancer. Gastroenterology. 2000 May;118(5):829-34. doi: 10.1016/s0016-5085(00)70168-5. PMID 10784581
- [Background] Engel C, Rahner N, Schulmann K, Holinski-Feder E, Goecke TO, Schackert HK, Kloor M, Steinke V, Vogelsang H, Moslein G, Gorgens H, Dechant S, von Knebel Doeberitz M, Ruschoff J, Friedrichs N, Buttner R, Loeffler M, Propping P, Schmiegel W; German HNPCC Consortium. Efficacy of annual colonoscopic surveillance in individuals with hereditary nonpolyposis colorectal cancer. Clin Gastroenterol Hepatol. 2010 Feb;8(2):174-82. doi: 10.1016/j.cgh.2009.10.003. Epub 2009 Oct 14. PMID 19835992
- [Background] Ahadova A, von Knebel Doeberitz M, Blaker H, Kloor M. CTNNB1-mutant colorectal carcinomas with immediate invasive growth: a model of interval cancers in Lynch syndrome. Fam Cancer. 2016 Oct;15(4):579-86. doi: 10.1007/s10689-016-9899-z. PMID 26960970
- [Background] Chambuso R, Kaambo E, Rebello G, Ramesar R. Correspondence on "Cancer risks by gene, age, and gender in 6350 carriers of pathogenic mismatch repair variants: findings from the Prospective Lynch Syndrome Database" by Dominguez-Valentin et al. Genet Med. 2022 May;24(5):1148-1150. doi: 10.1016/j.gim.2022.01.006. Epub 2022 Feb 12. No abstract available. PMID 35168886
- [Background] Lu KH, Wood ME, Daniels M, Burke C, Ford J, Kauff ND, Kohlmann W, Lindor NM, Mulvey TM, Robinson L, Rubinstein WS, Stoffel EM, Snyder C, Syngal S, Merrill JK, Wollins DS, Hughes KS; American Society of Clinical Oncology. American Society of Clinical Oncology Expert Statement: collection and use of a cancer family history for oncology providers. J Clin Oncol. 2014 Mar 10;32(8):833-40. doi: 10.1200/JCO.2013.50.9257. Epub 2014 Feb 3. No abstract available. PMID 24493721
- [Background] Kumar S, Dudzik CM, Reed M, Long JM, Wangensteen KJ, Katona BW. Upper Endoscopic Surveillance in Lynch Syndrome Detects Gastric and Duodenal Adenocarcinomas. Cancer Prev Res (Phila). 2020 Dec;13(12):1047-1054. doi: 10.1158/1940-6207.CAPR-20-0269. Epub 2020 Aug 28. PMID 32859614
- [Background] Capelle LG, Van Grieken NC, Lingsma HF, Steyerberg EW, Klokman WJ, Bruno MJ, Vasen HF, Kuipers EJ. Risk and epidemiological time trends of gastric cancer in Lynch syndrome carriers in the Netherlands. Gastroenterology. 2010 Feb;138(2):487-92. doi: 10.1053/j.gastro.2009.10.051. Epub 2009 Nov 10. PMID 19900449
- [Background] Kloor M, Huth C, Voigt AY, Benner A, Schirmacher P, von Knebel Doeberitz M, Blaker H. Prevalence of mismatch repair-deficient crypt foci in Lynch syndrome: a pathological study. Lancet Oncol. 2012 Jun;13(6):598-606. doi: 10.1016/S1470-2045(12)70109-2. Epub 2012 May 1. PMID 22552011
- [Background] Giorgi Rossi P, Vicentini M, Sacchettini C, Di Felice E, Caroli S, Ferrari F, Mangone L, Pezzarossi A, Roncaglia F, Campari C, Sassatelli R, Sacchero R, Sereni G, Paterlini L, Zappa M. Impact of Screening Program on Incidence of Colorectal Cancer: A Cohort Study in Italy. Am J Gastroenterol. 2015 Sep;110(9):1359-66. doi: 10.1038/ajg.2015.240. Epub 2015 Aug 25. PMID 26303133
- [Background] Ladabaum U, Ford JM, Martel M, Barkun AN. American Gastroenterological Association Technical Review on the Diagnosis and Management of Lynch Syndrome. Gastroenterology. 2015 Sep;149(3):783-813.e20. doi: 10.1053/j.gastro.2015.07.037. Epub 2015 Jul 27. No abstract available. PMID 26226576
- [Background] Kalady MF, Kravochuck SE, Heald B, Burke CA, Church JM. Defining the adenoma burden in lynch syndrome. Dis Colon Rectum. 2015 Apr;58(4):388-92. doi: 10.1097/DCR.0000000000000333. PMID 25751794
- [Background] Schwitalle Y, Kloor M, Eiermann S, Linnebacher M, Kienle P, Knaebel HP, Tariverdian M, Benner A, von Knebel Doeberitz M. Immune response against frameshift-induced neopeptides in HNPCC patients and healthy HNPCC mutation carriers. Gastroenterology. 2008 Apr;134(4):988-97. doi: 10.1053/j.gastro.2008.01.015. Epub 2008 Jan 11. PMID 18395080
- [Background] Saeterdal I, Bjorheim J, Lislerud K, Gjertsen MK, Bukholm IK, Olsen OC, Nesland JM, Eriksen JA, Moller M, Lindblom A, Gaudernack G. Frameshift-mutation-derived peptides as tumor-specific antigens in inherited and spontaneous colorectal cancer. Proc Natl Acad Sci U S A. 2001 Nov 6;98(23):13255-60. doi: 10.1073/pnas.231326898. Epub 2001 Oct 30. PMID 11687624
- [Background] Linnebacher M, Gebert J, Rudy W, Woerner S, Yuan YP, Bork P, von Knebel Doeberitz M. Frameshift peptide-derived T-cell epitopes: a source of novel tumor-specific antigens. Int J Cancer. 2001 Jul 1;93(1):6-11. doi: 10.1002/ijc.1298. PMID 11391614
- [Background] Reuschenbach M, Kloor M, Morak M, Wentzensen N, Germann A, Garbe Y, Tariverdian M, Findeisen P, Neumaier M, Holinski-Feder E, von Knebel Doeberitz M. Serum antibodies against frameshift peptides in microsatellite unstable colorectal cancer patients with Lynch syndrome. Fam Cancer. 2010 Jun;9(2):173-9. doi: 10.1007/s10689-009-9307-z. PMID 19957108
- [Background] Kloor M, Reuschenbach M, Pauligk C, Karbach J, Rafiyan MR, Al-Batran SE, Tariverdian M, Jager E, von Knebel Doeberitz M. A Frameshift Peptide Neoantigen-Based Vaccine for Mismatch Repair-Deficient Cancers: A Phase I/IIa Clinical Trial. Clin Cancer Res. 2020 Sep 1;26(17):4503-4510. doi: 10.1158/1078-0432.CCR-19-3517. Epub 2020 Jun 15. PMID 32540851